CLINICAL TRIAL: NCT05835895
Title: A Phase 1b, Randomized, Double-Blinded, Placebo-Controlled Dose Ranging Study to Evaluate Safety, Tolerability and Pharmacodynamics of a Single Intra-articular Injection of GNSC-001 Gene Therapy in Subjects With Osteoarthritis of the Knee
Brief Title: Safety and Pharmacodynamics of GNSC-001 Intra-articular Injection for Knee Osteoarthritis
Acronym: DONATELLO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genascence Corporation (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPRO-22-001; CLIN2-14265 (Other Grant/Funding Number: California Institute for Regenerative Medicine)
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee; Osteo Arthritis Knee; Knee Osteoarthritis
Keywords: Gene therapy; Adeno-associated virus; Intra-articular; GNSC-001; Genascence; Knee pain; Knee arthritis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- GNSC-001 (low dose) (Experimental)
  Interventions: Genetic: GNSC-001
- GNSC-001 (low dose) + transient immune-modulation (oral) (Experimental)
  Interventions: Genetic: GNSC-001; Drug: transient immune-modulation
- GNSC-001 (high dose) (Experimental)
  Interventions: Genetic: GNSC-001
- GNSC-001 (high dose) + transient immune-modulation (oral) (Experimental)
  Interventions: Genetic: GNSC-001; Drug: transient immune-modulation
- GNSC-001 (high dose) + transient immune-modulation (oral + injectable) (Experimental)
  Interventions: Genetic: GNSC-001; Drug: transient immune-modulation
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: GNSC-001 — intra-articular injection
  Other Names: sc-rAAV2.5IL-1Ra
  Arms: GNSC-001 (high dose); GNSC-001 (high dose) + transient immune-modulation (oral + injectable); GNSC-001 (high dose) + transient immune-modulation (oral); GNSC-001 (low dose); GNSC-001 (low dose) + transient immune-modulation (oral)
Drug: transient immune-modulation — oral
  Arms: GNSC-001 (high dose) + transient immune-modulation (oral + injectable); GNSC-001 (high dose) + transient immune-modulation (oral); GNSC-001 (low dose) + transient immune-modulation (oral)
Drug: transient immune-modulation — intra-articular injection
  Arms: GNSC-001 (high dose) + transient immune-modulation (oral + injectable)
Drug: Placebo — intra-articular injection
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to determine if a single injection of 1 or more dose levels of adeno-associated virus (AAV) gene therapy (GNSC-001) is safe and tolerated compared to placebo in participants with painful osteoarthritis (OA) of the knee.

ELIGIBILITY:
Key Inclusion Criteria:

* OA in at least one knee (the 'target knee'), confirmed using centrally read X-ray with a Kellgren-Lawrence (KL) score of 2 or 3
* Western Ontario & McMaster University Osteoarthritis Index (WOMAC) pain score ≥ 20 (on a 50-point numerical rating scale) in the target knee during the seven days prior to Screening
* Persistent moderate to severe symptoms in the target knee, despite failure or intolerance of a 3-month trial of at least 2 conservative therapies (e.g., activity modification, weight loss, physical therapy, opioids, and anti-inflammatory medications, and injection of hyaluronic acid or steroids)
* Successful extraction of synovial fluid at Screening
* Negative pregnancy test at Screening and Baseline (subjects of childbearing potential [SOCBP])

Key Exclusion Criteria:

* Current or documented history of inflammatory arthritis (such as gout or rheumatoid arthritis), inflammation of connective tissue, or other immunological disease
* Any form of joint degeneration as part of another syndrome (e.g., Ehler's Danlos, Stickler syndrome, etc.)
* Surgery in the target knee within the 6 months prior to screening
* Previous partial or total joint replacement in target knee
* Significant and clinically evident malalignment of the target knee that would impact the subject's function, as determined by the Investigator
* Body mass index (BMI) > 38 kg/m2
* Clinically significant abnormal laboratory values at Screening in laboratory parameters that in the opinion of the Investigator, could represent a potential risk to participant safety:
* Plans to have, elective surgery of other joints or spine or intra-articular injections in the target knee, within the next 12 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Month 12
Severity of TEAEs and SAEs | Month 12

SECONDARY OUTCOMES:
Synovial fluid Interleukin-1 Receptor Antagonist (IL-1Ra) levels | Month 12
Synovial fluid Interleukin-1 Receptor Antagonist (IL-1Ra) levels | Months 1, 3, 6, and 24 months
Change in synovial Interleukin-1 Receptor Antagonist (IL-1Ra) levels over time | Baseline to Months 1, 3, 6, 12 and 24

OTHER OUTCOMES:
Immunogenicity of a single dose of GNSC-001 | Month 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jeymi Tambiah, MBChB, Study Director — Genascence Corporation
Locations (9):
- United States (9):
  - Alliance for Medical Research Mobile, Mobile, Alabama
  - Biosolutions Clinical Research Center, La Mesa, California
  - UC San Diego, San Diego, California
  - Well Pharma Medical Research, Miami, Florida
  - South Florida Research, Miami Springs, Florida
  - Premier Medical Associates, The Villages, Florida
  - Alliance for Multispecialty Research Kansas City, Kansas City, Missouri
  - West Clinical Research, Morehead City, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans CH, Ghivizzani SC, Robbins PD. Osteoarthritis Gene Therapy: A 30-Year Journey From Concept to Clinical Trials. J Orthop Res. 2026 Feb;44(2). doi: 10.1002/jor.70141. PMID 41607103
- [Derived] Chen L, Huang FL, Tang Q, Zhao ZK, Ye ZY, Liang JH. Targeted therapy for knee osteoarthritis: From basic to clinics. Medicine (Baltimore). 2025 Aug 15;104(33):e43686. doi: 10.1097/MD.0000000000043686. PMID 40826764
- [Derived] Evans CH, Ghivizzani SC, Robbins PD. The 2024 OREF Clinical Research Award: Progress Toward a Gene Therapy for Arthritis. J Am Acad Orthop Surg. 2024 Dec 1;32(23):1052-1060. doi: 10.5435/JAAOS-D-24-00831. Epub 2024 Oct 17. PMID 39284030